CLINICAL TRIAL: NCT07298655
Title: 3D Contrast Enhanced Microvascular Ultrasound of Carotid Atherosclerosis for the Detection of Carotid Plaque Neo-Revascularisation.
Acronym: Carotid Neo3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC/2024/001; 349094 (Other: IRAS)
Record Dates: First submitted 2025-11-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Carotid Atherosclerosis; Ultrasound; Plaque Neovascularization
Keywords: Carotid atherosclerosis; Carotid Ultrasound; Plaque Neovascularisation
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Intervention Model Description: prospective proof of concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D contrast enhanced microvascular carotid ultrasound (Experimental): Patients will be cannulated in order to allow infusion of SonoVue® (Bracco, Milan) microbubble contrast agent. A 5ml vial will be made up into an infusion and given at a rate to allow adequate arterial opacification according to standard clinical practices. Initial 2D B-mode ultrasound images will be taken of the carotid arteries using a standard 3- to 11- MHz linear transducer on an EPIC CVx machine (Philips Medical Systems). This will confirm the presence of plaque and allow a scouted location for the desired row-column array transducer images. CEUS images will be taken with the 2D matrix array probe to allow comparative baseline images. Once the desired area has been located and CEUS images have confirmed plaque, the row-column array probe, manipulated by a clinician, will be used to take the 3D images. Microbubble contrast infusion will be given followed by a scan with the row-column array transducer which should take 2-5 minutes, taking multiple acquisitions if required. A member
  Interventions: Diagnostic Test: 3D Contrast Enhanced Microvascular Carotid Ultrasound

INTERVENTIONS:
Diagnostic Test: 3D Contrast Enhanced Microvascular Carotid Ultrasound — Patients will be cannulated in order to allow infusion of SonoVue® (Bracco, Milan) microbubble contrast agent. A 5ml vial will be made up into an infusion and given at a rate to allow adequate arterial opacification according to standard clinical practices. Initial 2D B-mode ultrasound images will be taken of the carotid arteries using a standard 3- to 11- MHz linear transducer on an EPIC CVx machine (Philips Medical Systems). This will confirm the presence of plaque and allow a scouted location for the desired row-column array transducer images. CEUS images will be taken with the 2D matrix array probe to allow comparative baseline images. Once the desired area has been located and CEUS images have confirmed plaque, the row-column array probe, manipulated by a clinician, will be used to take the 3D images. Microbubble contrast infusion will be given followed by a scan with the row-column array transducer which should take 2-5 minutes, taking multiple acquisitions if required. A member

SUMMARY:
Atherosclerotic plaques, the build-up of fatty materials within our arteries, can develop over a long period of time without causing any symptoms.

These plaques may continue to grow and rupture causing narrowing and blockages of the blood vessels. This can lead to serious cardiovascular disease such as a heart attack or stroke causing over 160,000 deaths each year.

Lots of research has been done on why particular groups of people may develop atherosclerosis and controlling risk factors such as diabetes and high blood pressure go a long way to reduce people's risks. However, despite the treatments we have available and controlling these risk factors, some people unfortunately still go on to develop a potentially serious disease.

Further research has shown us that certain plaques in the blood vessels may be more vulnerable to rupturing compared to others. So far we know that plaques with thin caps, soft centres or those that are able to grow their own tiny blood vessels are more likely to rupture. We have now started to develop new imaging methods to try and help us detect these vulnerabilities. The hope is by being able to detect more vulnerable plaques we may be able to treat these earlier and therefore more effectively.

There are different scans available to try and visualise the tiny vessels within these plaques in the neck arteries. These include, MRI (a Magnetic Resonance Imaging scan, taking pictures using a small tunnel), CT (Computed Tomography, uses a ring-shaped machine to take pictures), and ultrasound. Ultrasound has the benefit of being free of ionising radiation and iodinated contrast, therefore posing less risk to patients. However, current ultrasound uses 2D ultrasound. Although this has shown promising results, our blood vessels and any plaques are 3D structures so we don't get to see the whole plaque using 2D imaging and therefore may miss important information. The available 3D probes in use at the moment are not able to visualise the tiny vessels accurately enough.

This study uses a different 3D ultrasound probe and ultrasound machine that is able to produce many more images than our usual probes. By taking images with this probe and using offline computer programmes to track the contrast through structures we hope that this system will be able to give us a visualisation of the whole plaque enabling us to detect any new blood vessels more accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old.
2. Previously consent for participation in the SECURE trial and have undergone carotid CEUS.
3. Found to have at least one carotid plaque present on carotid CEUS.
4. Able to give informed consent to participate in the study and its procedures.

Exclusion Criteria:

1. Age <18 years old.
2. Unable to provide informed consent to participate in the study and its procedures.
3. Allergy to microbubble contrast agents.
4. Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Detection of carotid plaque neovascularisation | Baseline
  Can the 3D row-column array transducer detect intra-plaque neovascularisation in carotid plaques comparable to 2D CEUS

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, MD, Principal Investigator — LNWH Trust
Locations (1):
- Northwick Park Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided